CLINICAL TRIAL: NCT03396510
Title: Electronic Symptom Monitoring Intervention for Hospitalized Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alliance for Clinical Trials in Oncology Cancer Control Program (CCP) (Unknown)
Responsible Party: Principal Investigator, Ryan Nipp, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-567
Record Dates: First submitted 2018-01-03; First posted 2018-01-11 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: Cancer Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMPROVED intervention (Experimental): Patients randomized to the IMPROVED intervention will self-report their symptoms each day using a tablet computer. If any patient refuses or is unable to complete the symptom assessment on the computer, the study team will permit them to use paper versions. At morning rounds each day, the clinical team will view reports detailing their patients' symptom burden. Patients randomized to IMPROVED will have their symptoms presented to their inpatient oncology team, but the study team will not provide guidance about what actions to take in response to patients' symptoms.
  Interventions: Other: IMPROVED intervention
- Usual Care (No Intervention): Usual Care per hospital standard will be administered. Participants receiving usual care will also self-report their symptoms each day using tablet computers. However, these patients' clinicians will not receive their symptom reports.

INTERVENTIONS:
Other: IMPROVED intervention — Patients randomized to IMPROVED will self-report their symptoms each day using a tablet computer. If any patient refuses or is unable to complete the symptom assessment on the computer, the investigators will permit them to use paper versions. At morning rounds each day, the clinical team will view reports detailing their patients' symptom burden. Patients randomized to IMPROVED will have their symptoms presented to their inpatient oncology team, but the investigators will not provide guidance about what actions to take in response to patients' symptoms.
  Arms: IMPROVED intervention

SUMMARY:
This research study is evaluating a new way to deliver oncology care for patients with cancer

DETAILED DESCRIPTION:
Patients with cancer may experience a considerable symptom burden, often requiring hospitalizations for symptom management. The study doctors want to know if daily electronic monitoring of the symptoms, such as pain, nausea, constipation, and diarrhea may improve care while participants are hospitalized.

The goal of this study is to evaluate a new way to deliver oncology care where patients' symptoms are systematically monitored during their hospital admission. The investigators are studying whether patients whose clinicians receive their patients' detailed symptom reports each day have improved symptom management compared to those whose clinicians do not receive their patients' detailed symptom reports each day.

The study will use questionnaires to measure the participant symptoms and involves participating in a study for as long as the participants are admitted to the hospital. The information the investigators collect will help them determine if electronic symptom monitoring improves the care of patients with cancer

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with advanced cancer (defined as receiving treatment with palliative intent as per chemotherapy order entry designation, oncology clinic notes, and/or trial consent forms, or not receiving chemotherapy but followed for incurable disease as per oncology clinic notes)
* Admitted to the oncology service at Massachusetts General Hospital
* Verbal fluency in English

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Admitted electively
* Participated during a previous admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of days with improved symptoms between study arms | 2 years
  Using ESAS and PHQ symptoms, the investigators will compare the proportion of days that symptoms improved in standard care versus IMPROVED.

SECONDARY OUTCOMES:
Proportion of days with worsened symptoms between study arms | 2 years
  Using ESAS and PHQ symptoms, the investigators will compare the proportion of days that symptoms worsened in standard care versus IMPROVED.
Change in patients' symptom scores from baseline to discharge | 2 years
  Using ESAS and PHQ symptoms, the investigators will compare the average change in symptom burden for patients in standard care versus IMPROVED.
Hospital length of stay (measured continuously as days admitted to the hospital) between study arms | 2 years
  The investigators will compare hospital length of stay (measured continuously as days admitted to the hospital) between study arms.
Hospital readmissions within 30 days of prior hospital discharge between study arms | 30 days
  The investigators will compare readmissions within 30 days of prior hospital discharge between study arms.
Hospital readmissions within 90 days of prior hospital discharge between study arms | 90 days
  The investigators will compare readmissions within 90 days of prior hospital discharge between study arms.

OTHER OUTCOMES:
Age as a moderator of the effect of IMPROVED on symptom burden | 2 years
  The investigators will explore age as a potential moderator on the effect of IMPROVED on symptom burden.
Age as a moderator of the effect of IMPROVED on hospital length of stay | 2 years
  The investigators will explore age as a potential moderator on the effect of IMPROVED on hospital length of stay.
Age as a moderator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore age as a potential moderator on the effect of IMPROVED on hospital readmissions.
Sex as a moderator of the effect of IMPROVED on symptom burden | 2 years
  The investigators will explore sex as a potential moderator on the effect of IMPROVED on symptom burden.
Sex as a moderator of the effect of IMPROVED on hospital length of stay | 2 years
  The investigators will explore sex as a potential moderator on the effect of IMPROVED on hospital length of stay.
Sex as a moderator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore sex as a potential moderator on the effect of IMPROVED on hospital readmissions.
Cancer type as a moderator of the effect of IMPROVED on symptom burden | 2 years
  The investigators will explore cancer type as a potential moderator on the effect of IMPROVED on symptom burden.
Cancer type as a moderator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore cancer type as a potential moderator on the effect of IMPROVED on hospital readmissions.
Cancer type as a moderator of the effect of IMPROVED on hospital length of stay | 2 years
  The investigators will explore cancer type as a potential moderator on the effect of IMPROVED on hospital length of stay.
Baseline symptom burden as a moderator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore baseline symptom burden as a potential moderator on the effect of IMPROVED on hospital readmissions.
Baseline symptom burden as a moderator of the effect of IMPROVED on hospital length of stay | 2 years
  The investigators will explore baseline symptom burden as a potential moderator on the effect of IMPROVED on hospital length of stay.
Baseline symptom burden as a moderator of the effect of IMPROVED on symptom burden | 2 years
  The investigators will explore baseline symptom burden as a potential moderator on the effect of IMPROVED on symptom burden.
Hospital length of stay as a moderator of the effect of IMPROVED on symptom burden | 2 years
  The investigators will explore hospital length of stay as a potential moderator on the effect of IMPROVED on symptom burden.
Hospital length of stay as a moderator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore hospital length of stay as a potential moderator on the effect of IMPROVED on hospital readmissions.
Symptom burden as a mediator of the effect of IMPROVED on hospital length of stay | 2 years
  The investigators will explore whether improvements in symptom burden mediate the benefit of the intervention on hospital length of stay.
Symptom burden as a mediator of the effect of IMPROVED on hospital readmissions | 2 years
  The investigators will explore whether improvements in symptom burden mediate the benefit of the intervention on hospital readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nipp RD, Horick NK, Qian CL, Knight HP, Kaslow-Zieve ER, Azoba CC, Elyze M, Landay SL, Kay PS, Ryan DP, Jackson VA, Greer JA, El-Jawahri A, Temel JS. Effect of a Symptom Monitoring Intervention for Patients Hospitalized With Advanced Cancer: A Randomized Clinical Trial. JAMA Oncol. 2022 Apr 1;8(4):571-578. doi: 10.1001/jamaoncol.2021.7643. PMID 35142814